CLINICAL TRIAL: NCT00921466
Title: Pilot Study to Assess Feasibility, Reliability and Validity of the e-SSRS-IVR
Acronym: e-SSRS-IVR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rogers Center for Research & Training, Inc. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Dr John Greist, Rogers Center for Research and Training, Inc
Other Study IDs: 113235
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Evaluate the clinical content of the e-SSRS-IVR

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hospital Patients/Hospital Employees
- Hospital employees: A group of 10 hospital employees used as baseline

SUMMARY:
The proposed study is designed to evaluate the clinical contents of the e-SSRS-IVR with respect to 1.the intent of the instrument (assess face and content validity), 2. system validation with respect to programming integrity, 3. implementation feasibility in clinical ill and healthy patient populations, and 4. criterion/predictive validity to discriminate patient population with known clinical status differences.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults, able/willing to read and provide written consent

Exclusion Criteria:

* Dementia, delirium, psychosis or deafness.
* Control subjects will be excluded for any MINI lifetime MDD or dysthymia diagnosis of a DSM-IV disorder except for specific phobia or dependence on nicotine and caffeine.
* Inpatients not admitted with suicidal ideations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be recruited from a single clinical site (Rogers Memorial Hospital, Milwaukee WI). Half of the subjects will be recruited through public advertisement for Rogers Hospital employees and the other half will be recruited from recent inpatient psychiatric admissions.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John H Greist, MD, Principal Investigator — Rogers center for Research and Training, Inc
Locations (1):
- Rogers Center for Research and Training, Inc, Milwaukee, Wisconsin, United States

REFERENCES:
- See also: Related Info — http://rogershospital.org